CLINICAL TRIAL: NCT03452748
Title: Fourier Transformed Infrared Spectroscopy in Macular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of the department of Ophthalmology, principal investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FTIR
Record Dates: First submitted 2018-02-22; First posted 2018-03-02 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Epiretinal Membrane; Macular Hole
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations | interventions — Spectroscopy, Fourier Transform Infrared

STUDY DESIGN:
Intervention Model Description: all excised membranes will be examined with FTIR spectroscopy, there will be no control group
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FTIR arm (Experimental): all excised membranes are examined with FTIR spectroscopy
  Interventions: Device: FTIR spectroscopy

INTERVENTIONS:
Device: FTIR spectroscopy — FTIR spectroscopy examines collagen fibers in the excised membranes

SUMMARY:
Epiretinal membranes (ERM) are disorders leading to vision loss and metamorphopsia. Vitrectomy with membrane peeling has developed to be the gold-standard in treatment of ERM. ERM can be well visualized with spectral domain optical coherence tomography (SD-OCT).

The aim of the study is to examine ERM and internal limiting membranes (ILM) exzised during routine macular surgery with fourier transformed infrared spectroscopy (FTIR) and compare results to optic coherence tomography (OCT) findings.

DETAILED DESCRIPTION:
Purpose of the present study is to analyse components of ERM and ILM, giving hints for the origin of cells producing ERM. In contrast to electron microscopy, FTIR spectroscopy does not need any chemical fixation of the membranes and therefore structure of components of ERM and ILM are not changed by fixation.

In total, 20 eyes with idiopathic ERM, 10 eyes with lamellar macular hole, 10 eyes with full thickness macular hole and 10 eyes with diabetic ERM will be examined. To our knowledge there are no previous reports about FTIR spectroscopy of ERM and ILM, therefore the study will be performed as an exploratory pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic ERM, lamellar macular holes, full thickness macular holes, diabetic ERM and the indication for surgery (visual symptoms)
* Age 21 and older
* written informed consent for surgery and participation in the study prior to surgery

Exclusion Criteria: - Macular edema due to other reasons than ERM

* Hereditary macular disorders
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
collagen | 3 months
  occurrence of different types of collagen fibres in the excised membranes

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Principal Investigator — VIROS at Hanuschkrankenhaus
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria